CLINICAL TRIAL: NCT01672463
Title: Phase 1b Clinical Trial of IV OKN-007 in a Pilot Cohort of Human Recurrent Malignant Glioma Patients
Brief Title: Clinical Trial of IV OKN-007 in a Pilot Cohort of Human Recurrent Malignant Glioma Patients
Acronym: OKN-007
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oblato, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI57337
Record Dates: First submitted 2012-08-21; First posted 2012-08-24 (Estimated); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Recurrent Malignant Glioma
MeSH Terms: conditions — Glioma | interventions — OKN 007

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All patients (Experimental): All participants enrolled in this study
  Interventions: Drug: OKN-007

INTERVENTIONS:
Drug: OKN-007 — Dose escalation/PK cohort: 20 mg/kg, 40 mg/kg or 60 mg/kg OKN-007 via IV infusion, given 3x/week for the first 4 weeks, then 2x/week for the next 4 weeks, then 1x/week thereafter.
  Expansion cohort: MTD via IV infusion given 3x/week for the first 4 weeks, then 2x/week for the next 4 weeks, then 1x/week thereafter.

SUMMARY:
This is an open label Phase 1b clinical trial of IV administration of OKN-007 in a pilot cohort of human recurrent malignant glioma patients. All patients will have been previously treated with the standard-of-care treatment which includes surgical resection, radiation and chemotherapy, and in some cases treatment for recurrent disease with investigational agents or bevacizumab (Avastin). Patients with unequivocal recurrence (first or greater) established by MRI with and without contrast (e.g., Gd-DTPA (Gadolinium-diethylene triamine pentacetic acid) and meeting inclusion and exclusion criteria, will be eligible for OKN-007 treatment on this protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed histopathology of WHO grade III glioma or WHO grade IV GBM at primary diagnosis
2. Unequivocal radiographic evidence of tumor progression by MRI within 14 days prior to registration
3. Prior radiotherapy
4. Prior Temozolomide treatment
5. Last cytotoxic chemotherapy 28 or more days or biologic therapy treatment 14 or more days before study start (greater than or equal to 42 days if nitrosourea was administered)
6. Karnofsky performance status greater than or equal to 60%
7. Full recovery (< grade 1) from the toxic effects of any earlier intervention and a minimum of 28 days from the administration of any investigational agent
8. Adequate renal, liver and bone marrow function:

   * Leukocytes >3,000/mcL
   * Absolute neutrophil count >1,500/mcL
   * Platelets >100,000/mcL
   * Total bilirubin within normal limits
   * AST / ALT (SGPT) <2.5 x ULN
   * Creatinine within normal limits
9. Patients must be >_18 years of age

Exclusion Criteria:

1. Second primary malignancy (except adequately treated basal cell carcinoma of the skin). Patients who had another malignancy in the past, but have been free of active disease for more than 2 years, are eligible
2. Have received treatment within the last 28 days with a drug that has not received regulatory approval for any indication at the time of study entry
3. Serious concomitant systemic disorders (for example, active infection or abnormal electrocardiogram (ECG) indicative of cardiac disease) that, in the opinion of the investigator, would compromise the safety of the patient and his/her ability to complete the study
4. Patients with moderate or severe renal impairment (calculated creatinine clearance of < 60 mL/min)
5. Patients with sodium, potassium, or creatinine serum electrolytes > grade 2.
6. Patients with PT/PTT above the upper limit of normal
7. Screening ECG abnormality documented by the investigator as medically significant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2012-12 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Number of Adverse events per patient | 24 months
  The primary objective is to determine MTD, tolerance, and safety of OKN-007 in patients with recurrent GBM and anaplastic glioma.

SECONDARY OUTCOMES:
PK level in participants | 24 months
  To determine drug levels of OKN-007 in blood.
6 month progression-free survival | 24 months
  To determine radiographic response rate and 6 month Progression-Free Survival (PFS) of patients treated with OKN-007. PFS is defined as the time from first drug treatment until objective tumor progression or death.

CONTACTS AND LOCATIONS:
Overall Officials: James Battiste, MD, PhD, Principal Investigator — • Oklahoma University
Locations (1):
- Oklahoma University, Oklahoma City, Oklahoma, United States